CLINICAL TRIAL: NCT02828514
Title: Nasal Resonance Change After Endoscopic Endonasal Transsphenoidal Skull Base Surgery: Analysis of Quality of Voice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Pornthep Kasemsiri, Department of Otorhinolaryngology, Khon Kaen University
Other Study IDs: IN58314
Record Dates: First submitted 2016-07-02; First posted 2016-07-11 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Voice Quality; Endoscopic Pituitary Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine nasal resonance change after endoscopic endonasal transsphenoidal skull base surgery. Furthermore, the quality of voice is assessed, also.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent endoscopic endonasal transsphenoidal skull base surgery

Exclusion Criteria:

* Patients under 18 year
* Patients cannot following command including loss of conscious
* Patients cannot speak including patient on tracheostomy tube
* Patients who has nasal tumor, nasal polyp, sinusitis
* Patients who has cleft lip cleft palate or submucosal cleft
* Patients who underwent adenotonsillectomy or palatoplasty in same setting with endoscopic pituitary surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent endoscopic endonasal transsphenoidal skull base surgery
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Nasal resonance change after endoscopic endonasal transsphenoidal surgery which was assessed by computer speech lab | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Pornthep Kasemsiri, MD., Principal Investigator — Khon Kaen University
Locations (1):
- Khon Kaen University, Khon Kaen, Khon Kean, Thailand

REFERENCES:
- [Derived] Kasemsiri P, Duangthongphon P, Prathanee B, Thongrong C. Nasal resonance changes after endoscopic endonasal transsphenoidal skull base surgery: Analysis of voice quality. Laryngoscope Investig Otolaryngol. 2021 Nov 19;6(6):1275-1282. doi: 10.1002/lio2.701. eCollection 2021 Dec. PMID 34938862